CLINICAL TRIAL: NCT06594770
Title: Time of Treatment of Hall Technique Versus Atraumatic Restorative Technique in the Management of Carious Primary Molars: a Randomized Clinical Trial
Brief Title: Time of Treatment in HALL Technique Vs ART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Doaa Mohamed Khalil, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hall technique VS ART
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Healthy
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ART (Experimental)
  Interventions: Procedure: Atraumatic Restorative Treatment
- HALL technique (Active Comparator)
  Interventions: Procedure: Hall technique

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment — A sharp excavator will be used to remove soft demineralized carious tissue from the patient's primary molar 2-The molar will then be restored with capsulated Glass Ionomer in accordance to ART procedure.
  3-Each capsule will be mixed for ten seconds and used for restoring teeth isolated by cotton rolls.
  4-After the cement is cured, excess material will be removed with an excavator and a carver.
  5-The occlusion will be tested for interferences with carbon paper. A layer of varnish coat will be applied to the surface and light-cured for 20 seconds .
  Arms: ART
Procedure: Hall technique — The procedure involves assessing the occlusion, contact points, and tooth shape. If contact points are present, orthodontic separators will be placed between the primary molars to create space for crown fitting, with the child seated upright to maintain airway safety. After 3 to 5 days, the separators will be removed, and loose plaque and debris will be cleared.
  The correct crown size will be selected, ensuring it doesn't impinge on adjacent teeth, and will be filled with glass ionomer cement. The child will be instructed to bite down for two minutes to ensure proper seating. Excess cement will be removed, and contacts will be flossed. Any initial occlusal discrepancies are expected to resolve within weeks.
  Arms: HALL technique

SUMMARY:
The goal of this clinical trial is to assess the time of treatment of Hall Technique versus Atraumatic Restorative Technique in the management of carious primary molars. The main questions it aims to answer are:

* Does the Hall Technique provide a faster and pain-free treatment compared to ART?
* How do the outcomes of both techniques impact children's acceptance and behavior? Researchers will compare the Hall Technique, which uses preformed metal crowns without caries removal, to Atraumatic Restorative Treatment, which uses hand instruments to selectively remove carious tissue.

Participants will:

* Receive treatment using either the Hall Technique or ART in a single session.
* Attend follow-up visits to monitor the effectiveness and acceptance of the treatment.
* Complete assessments on their experience and comfort during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age: From 4 to 6 years.
* Caries in primary molars within enamel/dentin with vital pulp.
* Healthy children.
* Cooperative children

Exclusion Criteria:

* Presence of signs and symptoms of necrosis.
* Root caries.
* History of spontaneous pain.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
time of treatment | during the procedure
  Time will be measured from the start of the procedure till its end using digital chronometer as a device and minutes as a unit.

SECONDARY OUTCOMES:
Postoperative Pain and discomfort | immediately after the procedure , 3month ,6 month and 12 month
  Immediately after the treatment, any pain and discomfort experienced by the child will be recorded using the Face Pain Scale - revised (FPS-R), which has six numbered faces from 0 to10 The (FPS-R). Each child will be asked to mark the face that reflects her or his experienced pain during the treatment. There is no pain visible on this face [indicating the face on the far left]. As you move from left to right, the faces get progressively more painful until you reach this one, which is incredibly painful [indicating the face on the far right]. The (FPS-R) faces will be scored as 0-2-4-6-8-10.
Child behavior | during the procedure
  At the end of the treatment session, the dentist classifies the child's behavior during the treatment according to Venham Behavior Rating Scale is a reliable system for rating behavior of children in the dental setting. ratings will be scored as 0-1-2-3-4-5
Canine overbite: HT | preoperatively , immediately after the procedure , 3 month , 6 month, 12 month
  the canine overbite will be measured only for the hall technique group. The canine overbite will be measured before the procedure using a Boley Gauge, either on the same side or the opposite side if the canine is missing. After assessing tooth shape and occlusion, a stainless-steel crown (SSC) will be partially seated on the tooth with glass ionomer cement. The child will bite on a cotton roll to fully seat the crown, after which excess cement will be removed, and the overbite will be recorded immediately after treatment.
Child anxiety | during the procedure
  At the end of the treatment session, the dentist classifies the child's anxiety during the treatment according to Venham Anxiety Rating Scale is a reliable system for rating anxiety of children in the dental setting. ratings will be scored as 0-1-2-3-4-5